CLINICAL TRIAL: NCT01246440
Title: A Phase II of Intraperitoneal Catumaxomab as a Consolidation Therapy in Patients With Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma in Second or Third Complete Clinical Disease Remission
Brief Title: Catumaxomab as a Consolidation Therapy in Patients With Ovarian Cancer in Second or Third Clinical Disease Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: Neovii Biotech (Industry)
Responsible Party: Principal Investigator, Secretaría Técnica GEICO, Antonio Gonzalez (Chairman GEICO), Grupo Español de Investigación en Cáncer de Ovario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICO-1001; 2010-018478-19 (EudraCT Number)
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Catumaxomab (Experimental)
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — Catumaxomab: 4 intraperitoneal infusions of catumaxomab over 11 days administered in a period of 3 hours through an intraperitoneal catheter with the following dosage: 1) 10 µg on Day 0. 2) 20 µg on Day 3. 3) 50 µg on Day 7. 4) 200 µg on Day 10.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of catumaxomab as consolidation treatment in patients with epithelial ovarian cancer in second or third complete remission.

DETAILED DESCRIPTION:
Epithelial ovarian cancer is the most lethal malignant gynecological tumor and the fourth most common cause of death by cancer among women. The highest incidence rates are observed in Eastern and Northern Europe, and in the United Status. In Spain, 3,262 new cases were diagnosed in 2002, and the figure is expected to rise to 3,722 cases in 2015 (Globocan 2002, International Agency for Research on Cancer -IARC).

The majority of patients with ovarian cancer are diagnosed at an advanced stage, and are treated with maximum cytoreductive surgery followed by intraperitoneal and/or intravenous chemotherapy. What is considered standard chemotherapy consists of a platinum (carboplatin or cisplatin) combined with a taxane, usually paclitaxel (Ozols, 2003; Armstrong 2006). Although many patients respond to the initial treatment, the majority experience subsequent recurrence of the disease, which is why they need to be treated with successive salvage therapies in an attempt to control the disease until it is converted into totally refractory (Markman, 2004). Only 20-30% of patients can be cured with current treatments, which is why it is necessary to investigate and develop new treatments and/or treatment strategies (Yap, 2009).

Although with the initial treatment based on cytoreductive surgery and platinum-based chemotherapy the large majority of patients achieve complete remission of the disease, 90% of the patients with sub-optimum cytoreductive surgery and 70% with optimum cytoreductive surgery develop a recurrence in the first 24 months. One of the treatment strategies being investigated to try and improve the results is the administration of consolidation or maintenance treatment to those patients that have achieved a complete response of their disease to reduce the risk of subsequent recurrence (Sabbatini, 2006).

In the last few years, various studies have established that investigating a possible therapeutic effect of consolidation or maintenance treatment following second or third complete clinical remission, obtained with a salvage chemotherapy, produces several advantages over the same strategy applied on a first complete clinical response: the median of progression-free survival after second or third complete response is shorter and more predictable -10 months-, and moreover the recurrence is practically universal (Markman 2004; Harrison, 2007; Levine, 2007; Markman, 2008; Juretza, 2008).

Catumaxomab has proven to be effective in patients with refractory tumours and recurring malignant ascites, i.e. patients with a very advanced disease, a large tumour and no treatment options. These clinical conditions are the worst for researching into any immune-based therapy, hence it seems logical to study the efficacy of catumaxomab in more favourable conditions.

Patients with ovarian cancer in second or third complete remission may be a more suitable population for investigating the intraperitoneal administration of catumaxomab as consolidation treatment: 1. 100% of the epithelial ovarian cancers express EpCAM (Epithelial cell adhesion molecule )(Kim, 2003; Bellone, 2009). 2. These patients present a minimal residual disease that cannot be eliminated with standard chemotherapy and is responsible for a subsequent recurrence in practically every patient, with a median progression-free survival of 10 months (Markman, 2004; Harrison, 2007). 3. The peritoneal cavity is a very common location for residual disease and/or recurrence in ovarian cancer (Ferrandina, 2006). 4. The absence of macroscopic disease in the peritoneal cavity may bring about a greater absorption of catumaxomab on the blood level, with a hypothetical greater efficacy on the systemic level without entailing a greater risk of toxicity (Heiss, 2008; Lordick, 2008).

The intention in this phase II study is to estimate the clinical benefit of consolidation treatment with catumaxomab in patients with epithelial ovarian cancer in second or third complete remission, by measuring progression-free survival, the percentage of progression-free patients at 12, 18 and 24 months, and comparing individually for each patient the duration of progression-free survival obtained following consolidation with catumaxomab with that observed in her first complete remission. If we observe a median of progression-free survival equal to or greater than 14 months, accompanied by a significant percentage of progression-free patients at 18 and 24 months, we will assess the possibility of subsequently designing a phase III study of consolidation with catumaxomab.

To improve the tolerability of catumaxomab, premedication will be administered with low-dose corticoids before each infusion of catumaxomab. The low doses of corticoids have been shown not to interfere with the efficacy of catumaxomab, but by reducing the release of certain cytokines like TNF-α (Tumor Necrosis Factor Alpha) they may reduce the associated adverse effects (Waltz, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent.
* Initial histopathologic diagnosis of epithelial ovarian cancer, cancer of the fallopian tube or primary peritoneal carcinoma
* Women ≥ 18 years
* ECOG performance status ≤ 1 (Eastern Cooperative Oncology Groupperformance)
* Initial surgical cytoreduction as primary treatment combinated with Platinum- based chemotherapy administered as part of primary therapy.

Failure of the primary treatment as manifested by recurrent disease that have achieved a second or third complete response with a second or third-line chemotherapy (platinum-based or not).

The complete response to the second or third-line chemotherapy is defined as non symptoms of cancer persistence, normal CA-125 (cancer antigen 125), negative medical examination, and no evidence of disease in a TAC.

* At least 4 cycles of second or third-line chemotherapy must have been administered
* Surgery performed at first or second relapse in conjunction with second or third-line chemotherapy is permitted.

Exclusion Criteria:

* Acute or chronic infection
* Concomitant treatment with cancer chemo- and/or radiotherapy
* Exposure to an investigational product within 28 days of first infusion
* Previous treatment with murine monoclonal antibodies
* Inadequate renal function: creatinine >1.5 upper limit of normal [ULN] and/ or calculated creatinine clearance ≥ 50 mL/min
* Inadequate hepatic function (AST, ALT, >2.5 xULN; bilirubin >1.5 xULN), Hypoalbuminaemia < 3 g/dL
* Platelets <80000 cells/mm3; absolute neutrophil count (ANC) <1000 cells/mm3,
* Hb < 8g/dL and PTT > 2 x ULN
* Patients with occlusive intestinal or symptomatic sub-occlusive intestinal within the last 30 days.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* Unable or unwilling to comply fully with the protocol.
* Any co-morbid disease that would increase risk of toxicity according to investigator judgment
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* Exposure to investigational product, cancer, chemo-or radiotherapy within the last 28 days (6 weeks for nitrosoureas or mitomycin C) before first infusion
* Known or suspected hypersensitivity to catumaxomab or similar antibodies
* Long-lasting steroid treatment (≥ 7 days), Patients should only be included after stepwise discontinuation and free of steroids for a minimum of 5 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  Progression-free survival per protocol is defined as the period from the commencement of the consolidation treatment (catumaxomab Day 0) and the recurrence of the disease or the last follow-up for the patients not developing a recurrence.

SECONDARY OUTCOMES:
Second progression-free survival (2PFS) | 3 years
  In patients in second complete remission, measured from the beginning of the treatment for the first recurrence until the date of the second recurrence of the disease, or the date of the last follow-up when the patient does not develop a recurrence of the disease.
Third progression-free survival (3PFS) | 3 years
  In patients in third complete remission, measured from the beginning of the treatment for the second recurrence until the date of the third recurrence of the disease, or the date of the last follow-up when the patient does not develop a recurrence of the disease.
Progression-free survival per protocol | 3 years
  Measured from the date of the beginning of the study treatment (catumaxomab Day 0) until the recurrence of the disease, or the date of the last follow-up when the patient does not develop a recurrence of the disease.
First progression-free survival | 3 years
  Which has to be recorded retrospectively, measured from the date of the initial treatment for the ovarian cancer (neoadjuvant chemotherapy or cytoreductive surgery) until the date of the first recurrence of the disease.
Duration of the treatment-free interval | 3 years
  Measured from the date of the administration of the last dose of catumaxomab until the date of the beginning of the following salvage treatment.
Overall survival rate | 3 years
  Measured from the date of the first administration of the study treatment (catumaxomab Day 0) until the death of the patient.
Incidence, intensity and causalidad of every adverse event. | 3 years
  The incidence, intensity and possible causality of every adverse event (AE). AEs will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 4.0.
Therapeutic compliance | 3 years
  Compliance and percentage of patients being given the 4th dose of catumaxomab in accordance with the treatment plan, Day 10.
The level of cells involved in the immune response | 3 years
  The level of cells involved in the immune response, including sub-populations of the T lymphocytes, B lymphocytes, "natural killer" cells, and antigen-processing cells measured in a sample of ovarian cancer (optional study)
Interval between the administration of the last dose of chemotherapy and the beginning of the treatment with catumaxomab | 3 years
  Interval between the administration of the last dose of chemotherapy and the beginning of the treatment with catumaxomab

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, Dra., Study Chair — Hospital de la Vall d'Hebron; Antonio Gonzalez, Dr., Study Chair — M.D. Anderson; Miguel Beltran, Dr., Principal Investigator — Institut Calatà d'Oncologia de Girona; Yolanda García, Dra., Principal Investigator — Corporació Sanitaria Parc Tauli; Andrés Póveda, Dr., Principal Investigator — Instituto Valenciano de Oncología; Ana Santaballa, Dra., Principal Investigator — Hospital Universitario La Fe de Valencia; Mª Elena García, Dra., Principal Investigator — Hospital José Maria Morales Meseguer; Andrés Redondo, Dr., Principal Investigator — Hospital Universitario La Paz; Ana Herrero, Dra., Principal Investigator — Hospital Miguel Servet; Juan Fernando Cuevas, Dr., Principal Investigator — Hospital Clínico Universitario de Santiago de Compostela; Arantxa Gonzalez, Dra., Principal Investigator — Hospital Son Dureta; Eva Guerra, Dra., Principal Investigator — Hospital Universitario Ramon y Cajal; Jesus García, Dr., Principal Investigator — Hospital Universitario Fundación Alcorcon; Jose Angel Arranz, Dr., Principal Investigator — Hospital Gregorio Marañon; Ana de Juan, Dra., Principal Investigator — Hospital Universitario de Valdecilla; Antonio Casado, Dr., Principal Investigator — Hospital San Carlos, Madrid; César Mendiola, Dr., Principal Investigator — Hospital Universitario 12 de Octubre
Locations (17):
- Spain (17):
  - Hospital de la Vall d'Hebron, Barcelona, Barcelona
  - Institut Català d'Oncologia de Girona, Girona, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Valdecilla, Santander, Cantabria
  - Hospital Universitario 12 de Octubre, Madrid, Madrdi
  - Hospital Universitario Fundación Alcorcon, Alcorcón, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - M.D. Anderson, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Son Dureta, Mallorca, Mallorca
  - Hospital Jose Maria Morales Meseguer, Murcia, Murcia
  - Hosptial Clinico Universitario de Santiago de Compostela, Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario La Fe de Valencia, Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza